CLINICAL TRIAL: NCT05743933
Title: Cohort Study of Adrenogenic Autonomic Cortisol Secretion
Status: Not yet recruiting | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Prof., Chongqing Medical University
Other Study IDs: AC-China 2023
Record Dates: First submitted 2023-02-16; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Diagnosis; Treatment; Adrenogenic Autonomic Cortisol Secretion
Keywords: Diagnosis and differential diagnosis; Treatment and prognosis; Adrenogenic Autonomic Cortisol Secretion
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Some subtye of disease should be diagnosed by DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Accidental adrenal tumor with 1mg-DST cortisol >50nmol/L
- Control group: Accidental adrenal tumor with 1mg-DST cortisol ≤50nmol/L

SUMMARY:
To investige the etiology, pathogenesis, diagnosis and treatment of adrenogenic autonomic cortisol secretion in Chinese adults.

DETAILED DESCRIPTION:
With the development of imaging detection technology and its wide application in clinic, the detection rate of adrenal incidentaloma (AI) has been greatly improved. In our previous study, 18.9% of AI were accompanied by autonomic cortisol secretion (ACS) in Chinese. The vast majority of ACS is mild (MACS). Due to the lack of typical Cushing manifestations and the low rate of progression to overt Cushing, MACS has received insufficient attention in the past. However, recent studies have found that MACS have a higher incidence of diabetes, hypertension, cardiovascular events, metabolic bone disease and mortality risk than those with non-functional adenomas. With appropriate treatment, the complications of MACS patients can be effectively improved. However, personalized treatment of MACS is a clinical difficulty. It is hard to determine whether the cortisol secretion of patients is caused by AI or whether patients will benifit from operation. There are some retrospective studies have provided some evidence, while prospective studies are lacking. The purpose of this study is to prospectively include patients with autonomic cortisol secretion, evaluate function and diagnosis, develop personalized treatment strategy, and follow up the prognosis. The research results will provide new evidence for standardized diagnosis and treatment of adrenogenic autonomic cortisol secretion in the future.

ELIGIBILITY:
Inclusion Criteria:

* CT examination revealed adrenal nodules (maximum diameter ≥10mm);
* Serum cortisol > 50nmol/L after 1mg dexamethasone inhibition test (1mg-DST).

Exclusion Criteria:

* Patients with primary aldosteronism (PA), pheochromocytoma, adrenal metastatic carcinoma, congenital adrenal hyperplasia (CAH), ganglionic neuroma/paraganglioma, schwannoma, adrenal hematoma and those with no definite diagnosis were evaluated by clinical and endocrine function.
* Patients with serious underlying diseases (such as liver and kidney failure, acute severe infection, etc.) that may affect the function of the hypothalamic-pituitary-adrenal axis (HPA axis); Pregnancy.
* Patients with a history of alcoholism, fatigue, trauma, infection, depression, glucocorticoid use, and other drugs affecting the function of the hypothalamic-pituitary-adrenal axis.
* Patients who are not willing to participate in and complete this study refuse to sign the written informed consent for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with adrenal incidentaloma and serum cortisol > 50nmol/L after 1mg dexamethasone inhibition test, without other situation mentioned in exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-17 (Estimated); Primary Completion 2033-02-15 (Estimated); Study Completion 2033-02-15 (Estimated)

PRIMARY OUTCOMES:
SUVmax value of PET-CT | 10 years
  To explore the value of 68[Ga]-Pentixafor PET-CT in the diagnosis of MACS

SECONDARY OUTCOMES:
Etiology and pathogenesis of adrenogenic autonomic cortisol secretion | 10 years
  To study the etiology and pathogenesis of adrenogenic autonomic cortisol secretion

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, PhD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jing Y, Hu J, Luo R, Mao Y, Luo Z, Zhang M, Yang J, Song Y, Feng Z, Wang Z, Cheng Q, Ma L, Yang Y, Zhong L, Du Z, Wang Y, Luo T, He W, Sun Y, Lv F, Li Q, Yang S. Prevalence and Characteristics of Adrenal Tumors in an Unselected Screening Population : A Cross-Sectional Study. Ann Intern Med. 2022 Oct;175(10):1383-1391. doi: 10.7326/M22-1619. Epub 2022 Sep 13. PMID 36095315
- [Result] Prete A, Subramanian A, Bancos I, Chortis V, Tsagarakis S, Lang K, Macech M, Delivanis DA, Pupovac ID, Reimondo G, Marina LV, Deutschbein T, Balomenaki M, O'Reilly MW, Gilligan LC, Jenkinson C, Bednarczuk T, Zhang CD, Dusek T, Diamantopoulos A, Asia M, Kondracka A, Li D, Masjkur JR, Quinkler M, Ueland GA, Dennedy MC, Beuschlein F, Tabarin A, Fassnacht M, Ivovic M, Terzolo M, Kastelan D, Young WF Jr, Manolopoulos KN, Ambroziak U, Vassiliadi DA, Taylor AE, Sitch AJ, Nirantharakumar K, Arlt W; ENSAT EURINE-ACT Investigators*; ENSAT EURINE-ACT Investigators. Cardiometabolic Disease Burden and Steroid Excretion in Benign Adrenal Tumors : A Cross-Sectional Multicenter Study. Ann Intern Med. 2022 Mar;175(3):325-334. doi: 10.7326/M21-1737. Epub 2022 Jan 4. PMID 34978855
- [Result] Deutschbein T, Reimondo G, Di Dalmazi G, Bancos I, Patrova J, Vassiliadi DA, Nekic AB, Debono M, Lardo P, Ceccato F, Petramala L, Prete A, Chiodini I, Ivovic M, Pazaitou-Panayiotou K, Alexandraki KI, Hanzu FA, Loli P, Yener S, Langton K, Spyroglou A, Kocjan T, Zacharieva S, Valdes N, Ambroziak U, Suzuki M, Detomas M, Puglisi S, Tucci L, Delivanis DA, Margaritopoulos D, Dusek T, Maggio R, Scaroni C, Concistre A, Ronchi CL, Altieri B, Mosconi C, Diamantopoulos A, Iniguez-Ariza NM, Vicennati V, Pia A, Kroiss M, Kaltsas G, Chrisoulidou A, Marina LV, Morelli V, Arlt W, Letizia C, Boscaro M, Stigliano A, Kastelan D, Tsagarakis S, Athimulam S, Pagotto U, Maeder U, Falhammar H, Newell-Price J, Terzolo M, Fassnacht M. Age-dependent and sex-dependent disparity in mortality in patients with adrenal incidentalomas and autonomous cortisol secretion: an international, retrospective, cohort study. Lancet Diabetes Endocrinol. 2022 Jul;10(7):499-508. doi: 10.1016/S2213-8587(22)00100-0. Epub 2022 May 6. PMID 35533704